CLINICAL TRIAL: NCT05524116
Title: Telehealth Exercise and Mindfulness for Pain in Osteoarthritis: A Feasibility Study
Brief Title: Telehealth Exercise and Mindfulness for Pain in Osteoarthritis
Acronym: TEMPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Responsible Party: Principal Investigator, Deepak Kumar, Assistant Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6492
Record Dates: First submitted 2022-08-25; First posted 2022-09-01 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
Keywords: telehealth; exercise; mindfulness; pain; feasibility
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity; Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Parallel-arm randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: For some of the outcomes that are not patient-reported, researchers collecting the at the post-intervention visit timepoint will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group TX (Telehealth Exercise) (Active Comparator): Participants in this group will receive a supervised and group-based exercise program once a week for 8 weeks via telehealth.
  Interventions: Behavioral: Exercise
- Group TMX (Telehealth Exercise and Mindfulness) (Experimental): Participants in this group will receive a supervised, group-based integrated mindfulness and exercise program once a week for 8 weeks via telehealth.
  Interventions: Behavioral: Mindful Exercise program

INTERVENTIONS:
Behavioral: Mindful Exercise program — In this 8-week intervention, components of Mindful Based Stress Reduction Program will be integrated with strengthening and neuromuscular exercises recommended for knee osteoarthritis. The goal of this program is to train participants how to be mindful during their exercises.
  Arms: Group TMX (Telehealth Exercise and Mindfulness)
Behavioral: Exercise — In this 8-week intervention, participants will be given recommended strengthening and neuromuscular exercises for knee osteoarthritis. Participants in both the intervention and control group will receive these exercises.
  Arms: Group TX (Telehealth Exercise)

SUMMARY:
This is a parallel-arm mixed-methods randomized controlled trial to investigate the feasibility of telehealth delivered mindful exercise vs. usual exercise interventions for people with knee osteoarthritis.

DETAILED DESCRIPTION:
In this RCT, the feasibility of an 8-week telehealth mindful exercise intervention compared to an 8-week telehealth exercise only intervention for people with knee osteoarthritis (OA) will be assessed. Forty adults with knee OA will be assigned to either a mindful exercise arm OR exercise arm. Both interventions will be delivered via real-time videoconferencing in a group setting (n=8-10 per group). All participants will be administered questionnaires for self-reported symptoms, mood, quality of life, etc. throughout the study period. Participants will be given the choice to opt in for in-person data collection visits wherein their physical function, muscle strength, sensitivity to painful stimuli, and brain function will be assessed before and at the end of the interventions. At the end of the 8-week interventions, 10 participants will be purposively sampled from each arm (n=20 total) for individual interviews to determine acceptability of the telehealth interventions. Feasibility of the intervention will be determined post-intervention by outcome measures such as recruitment rate, retention rate, and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Meet National Institute for Health and Clinical Excellence clinical guidelines for knee osteoarthritis (i.e., age ≥ 50 years, presence of activity related pain, presence of morning knee stiffness ≤ 30 minutes)
* BMI<40
* Knee pain on most days for 3 months or more
* Average overall knee pain severity of ≥= 4 on a 11-point numeric rating scale during previous week
* Able to attend remote sessions
* Can speak and understand English at a sufficient level to understand the study procedures and informed consent.
* Available for study duration

Exclusion Criteria:

* Contraindications to exercise
* Other pain in lower back or legs that is greater than knee pain
* Received physical therapy treatment for knee OA in the past 6 months or currently receiving physical therapy
* Received any mindfulness programs such as Tai Chi, meditation, etc. in the past 6 months or currently receiving such program
* Currently receiving chemotherapy or radiation therapy for cancer except non-melanoma skin cancer
* History of other disease that may involve the index joint including inflammatory joint disease such as rheumatoid arthritis, seronegative spondyloarthropathy (eg, ankylosing spondylitis, psoriatic arthritis, inflammatory bowel disease related arthropathy), crystalline disease (eg, gout or pseudogout), lupus erythematosus, knee joint infections, Paget's disease affecting the knee, or knee joint tumors.
* Any knee surgery in the previous 6 months
* Joint replacement in either hip or ankle
* Previous knee osteotomy partial or total knee replacement in either knee
* Planned major treatment for knee OA (e.g., surgery, injections, physical therapy) during the study period
* Planned major surgery in the next 6 months
* Corticosteroid or hyaluronic acid injections in either knee in the previous 3 months
* Neurological conditions that impacts motor functioning (e.g., stroke, Parkinson's disease, Alzheimer's disease, Multiple Sclerosis, diabetic neuropathy, etc).
* Pregnancy (self-report)
* Participation in another clinical trial for any joint or muscle pain
* Suspected or known drugs or alcohol abuse

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-10-04 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Kumar, PT, PhD, Principal Investigator — Boston University
Locations (1):
- Movement and Applied Imaging Lab, Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Requests will be considered on an individual basis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 45 participants were enrolled (i.e., signed the consent form) and 40 of these were randomized to Group TX (n=19) or Group TMX (n=21).
  Five participants withdrew from the study prior to randomization due to work schedule changes (n=2), severe back pain (n=1), family emergency (n=1), and lack of motivation (n=1).
Period: Baseline to Postintervention (Week 8)
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Started | 19 | 21
Completed | 19 | 18
Not Completed | 0 | 3
Not completed — Brain tumor flare up | 0 | 1
Not completed — concussion | 0 | 1
Not completed — hernia surgery | 0 | 1
Period: Week 8 to Follow-up (Week 14)
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Started | 19 | 18
Completed | 18 | 17
Not Completed | 1 | 1
Not completed — Caregiver for sick family member | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness) | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (7.4) | 63.8 (8.9) | 65.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Education [Count of Participants; unit: Participants]
  High school or College 1 - 3 years | 6 | 8 | 14
  Undergraduate, graduate, or doctorate | 13 | 13 | 26
Annual income [Count of Participants; unit: Participants]
  More than 50,000$ | 10 | 11 | 21
  Less than 50,000$ | 8 | 9 | 17
  Did not report | 1 | 1 | 2
Marital Status [Count of Participants; unit: Participants]
  Married | 9 | 10 | 19
  Widowed, divorced, single, or not reported | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Recruitment
Description: Number of participants that are randomized for the study
Time Frame: through the recruitment process, up to 6 months from the start of the study
Population: A total of 40 randomized over 6 months (Oct 2022 - March 2023)
Measure: Count of Participants; unit: Participants
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
Participants | 19 | 21

2. Primary Outcome: Attendance
Description: Proportion of sessions attended
Time Frame: post-intervention (at 8-weeks)
Measure: Mean (Standard Deviation); unit: % sessions attended
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
% sessions attended | 68 (34) | 54 (39)

3. Primary Outcome: Retention Rate
Description: Proportion of participants who complete patient-reported outcome surveys
Time Frame: post-intervention visit (at the end of 8-weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
Participants | 19 | 18

4. Primary Outcome: Participant Feedback Survey
Description: Custom scale measuring feedback on interventionists and interventions. Scores range from 0-4 (0 - Strongly Disagree, 1 - Disagree, 2 - Neither Agree no Disagree, 3 - Agree, and 4 - Strongly Agree)
Time Frame: 8-week
Population: On the 19 participants randomized to TX group, 18 provided data for this outcome at week 8. Of the 21 participants assigned to the TMX group, 17 provided data for this outcome at week 8.
  Since the TX group did not receive any mindfulness training, outcome related to rating of the mindfulness intervention or instructor were not collected for this group.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 18 | 17
score on a scale
  The exercise instructor demonstrated good knowledge | 3.56 [2 to 4] | 3.29 [2 to 4]
  The exercise instructor was a good role model | 3.44 [2 to 4] | 3.35 [2 to 4]
  The exercise instructor explained lessons clearly | 3.33 [1 to 4] | 3.38 [2 to 4]
  The exercise instructor was engaging | 3.39 [2 to 4] | 3.44 [2 to 4]
  The exercise instructor was helpful/answered all questions | 3.33 [1 to 4] | 3.44 [2 to 4]
  I enjoyed the exercise lessons | 3.11 [1 to 4] | 2.88 [1 to 4]
  I was engaged in the exercise lessons | 3.39 [1 to 4] | 3.12 [2 to 4]
  I was able to understand the exercise lessons | 3.56 [2 to 4] | 3.24 [2 to 4]
  I was able to integrate the information from the different exercise lessons | 3.39 [2 to 4] | 3.19 [2 to 4]
  I will be able to use the exercise lessons in my life | 3.22 [0 to 4] | 3.25 [2 to 4]
  The mindfulness instructor demonstrated good knowledge: number analyzed (Participants) | 0 | 17
  The mindfulness instructor demonstrated good knowledge |  | 3.35 [2 to 4]
  The mindfulness instructor was a good role model: number analyzed (Participants) | 0 | 17
  The mindfulness instructor was a good role model |  | 3.35 [2 to 4]
  The mindfulness instructor explained lessons clearly: number analyzed (Participants) | 0 | 17
  The mindfulness instructor explained lessons clearly |  | 3.24 [2 to 4]
  The mindfulness instructor was engaging: number analyzed (Participants) | 0 | 17
  The mindfulness instructor was engaging |  | 3.29 [2 to 4]
  The mindfulness instructor was helpful/answered all questions: number analyzed (Participants) | 0 | 17
  The mindfulness instructor was helpful/answered all questions |  | 3.29 [2 to 4]
  I enjoyed the mindfulness lessons: number analyzed (Participants) | 0 | 17
  I enjoyed the mindfulness lessons |  | 2.71 [1 to 4]
  I was engaged in the mindfulness lessons: number analyzed (Participants) | 0 | 17
  I was engaged in the mindfulness lessons |  | 3.12 [2 to 4]
  I was able to understand the mindfulness lessons: number analyzed (Participants) | 0 | 17
  I was able to understand the mindfulness lessons |  | 3.12 [1 to 4]
  I was able to integrate the information from the different mindfulness lessons: number analyzed (Participants) | 0 | 17
  I was able to integrate the information from the different mindfulness lessons |  | 3.24 [2 to 4]
  I will be able to use the mindfulness lessons in my life: number analyzed (Participants) | 0 | 17
  I will be able to use the mindfulness lessons in my life |  | 3 [2 to 4]

5. Primary Outcome: Satisfaction Scale
Description: Custom 4-item (0-10 scale) to determine satisfaction with individual components of the intervention (i.e.,, exercise, mindfulness, telehealth, and overall satisfaction). There are 4 items and each item is scored separately. Higher scores for each item mean greater satisfaction for that dimension.
Time Frame: 8-week
Population: On the 19 participants randomized to TX group, 18 provided data for this outcome at week 8. Of the 21 participants assigned to the TMX group, 17 provided data for this outcome at week 8.
  TX group did not receive the mindfulness intervention so the mindfulness item on this scale was not administered to this group
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 18 | 17
score on a scale
  Exercise component | 8.1 [2.0 to 10.0] | 8.2 [5.0 to 10.0]
  Mindfulness Component: number analyzed (Participants) | 0 | 17
  Mindfulness Component |  | 7.3 [2.0 to 10.0]
  Telehealth component | 8.1 [1.0 to 10.0] | 7.9 [5.0 to 10.0]
  General participation | 7.9 [1.0 to 10.0] | 8.1 [5.0 to 10.0]

6. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score
Description: Patient-reported outcome for knee pain and disability; a percentage score from 0 to 100, 0 representing extreme problems and 100 representing no problems.
Time Frame: baseline, 8-week, 14-week
Population: On the 19 participants randomized to TX group, 18 provided data for this outcome at week 8 and week 14. Of the 21 participants assigned to the TMX group, 17 provided data for this outcome at week 8 and week 14.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Pain Baseline | 61.3 [57.6 to 64.9] | 57.7 [52.6 to 62.7]
  Pain Week-8: number analyzed (Participants) | 18 | 17
  Pain Week-8 | 63.7 [57.9 to 69.5] | 61.8 [54.4 to 69.1]
  Pain Week-14: number analyzed (Participants) | 18 | 17
  Pain Week-14 | 63.8 [57.3 to 70.3] | 64.2 [57 to 71.4]
  Symptoms Baseline | 59.7 [54.3 to 65] | 59.4 [53.9 to 65]
  Symptoms Week-8: number analyzed (Participants) | 18 | 17
  Symptoms Week-8 | 63.1 [58.5 to 67.8] | 59.9 [53.7 to 66.1]
  Symptoms Week-14: number analyzed (Participants) | 18 | 17
  Symptoms Week-14 | 68.8 [63 to 74.5] | 62.1 [54 to 70.3]
  Activity of Daily Living Baseline | 72.1 [66.7 to 77.6] | 63 [57.8 to 68.1]
  Activity of Daily Living Week-8: number analyzed (Participants) | 18 | 17
  Activity of Daily Living Week-8 | 72.6 [66.4 to 78.8] | 68.2 [60.3 to 76.1]
  Activity of Daily Living Week-14: number analyzed (Participants) | 18 | 17
  Activity of Daily Living Week-14 | 71.4 [64.2 to 78.7] | 68.5 [62.4 to 74.6]
  Sports and Recreation Baseline | 48.1 [37.5 to 58.6] | 37.4 [31.1 to 43.7]
  Sports and Recreation Week-8: number analyzed (Participants) | 18 | 17
  Sports and Recreation Week-8 | 47.2 [34.2 to 60.3] | 40.6 [32.4 to 48.7]
  Sports and Recreation Week-14: number analyzed (Participants) | 18 | 17
  Sports and Recreation Week-14 | 42.8 [30.6 to 55.1] | 45.3 [36.5 to 54.1]
  Quality Of Life Baseline | 45.8 [41.6 to 50] | 41.1 [35.1 to 47.1]
  Quality Of Life Week-8: number analyzed (Participants) | 18 | 17
  Quality Of Life Week-8 | 49 [44.1 to 53.8] | 48.5 [42.4 to 54.6]
  Quality Of Life Week-14: number analyzed (Participants) | 18 | 17
  Quality Of Life Week-14 | 52.1 [46.4 to 57.8] | 52.6 [44.4 to 60.7]

7. Secondary Outcome: Pain, Enjoyment, General Activity Scale
Description: Assesses Pain Intensity and Interference. the response range is 0-10; the PEG scale score is the mean of the three individual item scores. Higher scores represent worse pain.
Time Frame: baseline, 8-week, 14-week
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Baseline | 4.9 [4.2 to 5.6] | 5.4 [4.6 to 6.1]
  Week-8: number analyzed (Participants) | 18 | 17
  Week-8 | 4 [2.9 to 5] | 3.9 [3 to 4.7]
  Week-14: number analyzed (Participants) | 18 | 17
  Week-14 | 3.9 [2.9 to 4.9] | 3.4 [2.5 to 4.4]

8. Secondary Outcome: Numeric Rating Scale - Nominated Activity
Description: average rating of knee pain from 0-10, where 0 represents no pain and 10 represents worst pain imaginable, in the past week in a nominated activity selected at baseline
Time Frame: baseline, 8-week, 14-week
Population: as for outcome 6
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Baseline | 6.1 [5.3 to 6.9] | 6.5 [6.1 to 6.9]
  Week-8: number analyzed (Participants) | 18 | 17
  Week-8 | 5.1 [4 to 6.2] | 5.2 [4.4 to 5.9]
  Week-14: number analyzed (Participants) | 18 | 17
  Week-14 | 4.8 [3.8 to 5.9] | 4.8 [3.8 to 5.7]

9. Secondary Outcome: Participant Global Impression of Change
Description: participant's rating of change in condition on a 14-point scale ranging from "a very great deal worse" to "a very great deal better". Values range from -7 to +7 (excluding 0). Score >=1 represent improvement and scores <= -1 represent worsening.
Time Frame: 8-week, 14-week
Population: On the 19 participants randomized to TX group, 18 provided data for this outcome at week 8 and week 14. Of the 21 participants assigned to the TMX group, 16 provided data for this outcome at week 8 and 17 provided data for this outcome at week 14.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 18 | 17
score on a scale
  Week-8: number analyzed (Participants) | 18 | 16
  Week-8 | 2.2 [1 to 3.4] | 2.4 [1.2 to 3.7]
  Week-14 | 1.4 [0.1 to 2.7] | 2.2 [1.1 to 3.3]

10. Secondary Outcome: Patient Global Assessment of Osteoarthritis
Description: participant's assessment of impact of osteoarthritis on their general health on a 0-100 mm scale. higher scores represent higher impact of disease or worse global health
Time Frame: baseline, 8-week, 14-week
Population: One participant in TX group and four participants in TMX Group were lost to follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Baseline | 59.8 [49.2 to 70.4] | 63.7 [54.7 to 72.6]
  Week-8: number analyzed (Participants) | 18 | 17
  Week-8 | 64.5 [54.5 to 74.5] | 65.7 [56.9 to 74.5]
  Week-14: number analyzed (Participants) | 18 | 17
  Week-14 | 60.2 [50.8 to 69.5] | 68.7 [60.7 to 76.7]

11. Secondary Outcome: Pain Catastrophizing Scale
Description: 3-item scale which measures of catastrophizing related to pain. Each item is rated on a 5-point scale: 0 (Not at all) to 4 (all the time).
Time Frame: baseline, 8-week
Population: On the 19 participants randomized to TX group, 18 provided data for this outcome at week 8. Of the 21 participants assigned to the TMX group, 17 provided data for this outcome at week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Baseline | 3.5 [2.7 to 4.4] | 3.9 [2.9 to 4.9]
  Week-8: number analyzed (Participants) | 18 | 17
  Week-8 | 3.4 [2.3 to 4.6] | 3.1 [2 to 4.1]

12. Secondary Outcome: Widespread Pain Index Symptom Severity Scale
Description: self-report on severity of cognitive symptoms such as fatigue, trouble thinking or remembering, waking up tired, and other physical symptoms such as headache, dizziness, etc. Each symptom is scored on a 4-point scale where 0 indicates no problem and 3 indicates severe problem. Scores are calculated by summing items, with higher scores (out of a maximum score of 12) indicating greater symptom severity.
Time Frame: baseline, 8-week
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 18 | 21
score on a scale
  Baseline | 3.9 [3 to 4.8] | 3.1 [2.2 to 4.1]
  Week-8: number analyzed (Participants) | 18 | 17
  Week-8 | 4.1 [2.9 to 5.3] | 3.7 [2.6 to 4.9]

13. Secondary Outcome: Pain DETECT
Description: self-report measure on presence of neuropathic pain. each question is scored from 0 to 5 where higher scores indicate higher gradation of pain. The final score is between -1 and 38 and a score of 19 and higher indicates higher likelihood of neuropathic pain
Time Frame: baseline, 8-week
Population: On the 19 participants randomized to TX group, 18 provided data for this outcome at week 8. Of the 21 participants assigned to the TMX group, 20 provided data at baseline and 16 provided data for this outcome at week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 18 | 20
score on a scale
  Baseline | 9.8 [7.1 to 12.4] | 8.5 [6.6 to 10.4]
  Week-8: number analyzed (Participants) | 18 | 16
  Week-8 | 9.4 [7 to 11.8] | 7.6 [4.9 to 10.4]

14. Secondary Outcome: Patient Health Questionnaire 8-item
Description: 8-item questionnaire assessing depression symptoms. Each question is scored from 0 to 3 where higher scores indicate higher frequency of experiencing depressive symptoms. Total score is the sum of individual item scores. Score range is 0-24. Higher total scores indicate greater severity of depression
Time Frame: baseline, 8-week, 14-week
Population: On the 19 participants randomized to TX group, 18 provided data for this outcome at week 14. Of the 21 participants assigned to the TMX group, 17 provided data for this outcome at week 8 and week 14.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Baseline | 4.6 [2.3 to 6.9] | 3 [1.7 to 4.3]
  Week-8: number analyzed (Participants) | 19 | 17
  Week-8 | 3.7 [2.2 to 5.3] | 3.9 [1.9 to 6]
  Week-14: number analyzed (Participants) | 18 | 17
  Week-14 | 3.9 [2.4 to 5.5] | 4.1 [1.9 to 6.3]

15. Secondary Outcome: Cognitive and Affective Mindfulness Scale - Revised
Description: 12-item scale on dispositional mindfulness. Items are rated on a 4-point Likert scale from 1 (rarely/not at all) to 4 (almost always). Scores on the scale are summed. Higher scores reflect greater mindfulness.
Time Frame: baseline, 8-week, 14-week
Population: On the 19 participants randomized to TX group, 18 provided data for this outcome at week 8 and 17 provided data at week 14. Of the 21 participants assigned to the TMX group, 17 provided data for this outcome at week 8 and week 14.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Baseline | 35.3 [32.7 to 37.8] | 37.4 [34.5 to 40.3]
  Week-8: number analyzed (Participants) | 18 | 17
  Week-8 | 33.9 [30.6 to 37.3] | 36.4 [33 to 39.9]
  Week-14: number analyzed (Participants) | 17 | 17
  Week-14 | 35.2 [32.1 to 38.4] | 37.3 [33.4 to 41.2]

16. Secondary Outcome: Fear Avoidance Beliefs Questionnaire - Physical Activity
Description: 4-item questionnaire to determine how one's fear avoidance beliefs contributes to the cognitive/affective part of their knee pain. Each item is scored from 0 to 6. Total scores are summation of each item scores. Range is 0-24. Higher total scores indicate greater fear of physical activity
Time Frame: baseline, 8-week
Population: as for outcome 11
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Baseline | 18.3 [16.1 to 20.5] | 15.5 [12.9 to 18.1]
  Week-8: number analyzed (Participants) | 18 | 17
  Week-8 | 16.7 [13.4 to 20] | 14.8 [11.6 to 18.1]

17. Secondary Outcome: Arthritis Self Efficacy Scale
Description: Questionnaire to assess confidence in one's capacity to function despite pain. Each item in the questionnaire is scored on a 1-10 scale. It provides three subscales of pain, function, and other symptoms calculated as average of items contributing to that subscale. Range for each subscale is 1-10. Higher scores indicate greater self-efficacy to manage osteoarthritis.
Time Frame: baseline, 8-week
Population: Of the 21 participants assigned to the TMX group, 16 provided data for this outcome at week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Pain Baseline | 6.5 [5.8 to 7.3] | 6.1 [5.6 to 6.6]
  Pain Week-8: number analyzed (Participants) | 19 | 16
  Pain Week-8 | 7.1 [6.3 to 7.9] | 6.2 [5.3 to 7.1]
  Function Baseline | 8 [7.4 to 8.7] | 7.7 [7.1 to 8.2]
  Function Week-8: number analyzed (Participants) | 19 | 16
  Function Week-8 | 8.1 [7.2 to 9.1] | 8 [7.2 to 8.8]
  Other symptoms Baseline | 7 [6.2 to 7.7] | 6.8 [6.2 to 7.3]
  Other symptoms Week-8: number analyzed (Participants) | 19 | 16
  Other symptoms Week-8 | 7.1 [6.3 to 7.9] | 7.2 [6.4 to 8.1]

18. Secondary Outcome: Chronic Pain Self-efficacy Questionnaire
Description: Measures three domains of pain self-efficacy: pain management, physical functioning, and coping with symptoms. Each item is scored on a scale of 0 (very uncertain) to 100 (very certain). Score for each domain is the average of all items contributing to that domain. Higher total scores indicate greater self-efficacy to manage one's chronic pain.
Time Frame: baseline, 8-week
Population: On the 19 participants randomized to TX group, 17 provided data for this outcome at week 8. Of the 21 participants assigned to the TMX group, 16 provided data for this outcome at week 8.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
Number analyzed (Participants) | 19 | 21
score on a scale
  Pain Baseline | 71.5 [64.6 to 78.4] | 66.2 [59.6 to 72.7]
  Pain Week-8: number analyzed (Participants) | 17 | 16
  Pain Week-8 | 66.8 [56.8 to 76.8] | 66.9 [59.1 to 74.8]
  Function Baseline | 86 [78.8 to 93.2] | 81.4 [74.7 to 88.1]
  Function Week-8: number analyzed (Participants) | 17 | 16
  Function Week-8 | 82.2 [72.3 to 92.2] | 78.2 [66.5 to 89.9]
  Coping Baseline | 68.1 [60.1 to 76] | 72.6 [66.3 to 78.8]
  Coping Week-8: number analyzed (Participants) | 17 | 16
  Coping Week-8 | 71.2 [62.1 to 80.3] | 70.5 [60.6 to 80.5]

19. Other Pre Specified Outcome: Arthritis - Rapid Estimate of Adult Literacy in Medicine (A-REALM)
Description: 66-word recognition adult health literacy test. Each correct pronunciation of word is scored as 1. The total score is classified into 1 to 4 reading grade levels where higher scores (61-66) represent ninth grade and above reading level
Time Frame: baseline
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Sit to Stand Test [OPTIONAL IN-PERSON VISIT]
Description: functional test that measures the time taken to sit and stand from chair five times
Time Frame: baseline, 8-week
Reporting Status: Not Posted

21. Other Pre Specified Outcome: 6-minute Walk Test [OPTIONAL IN-PERSON VISIT]
Description: functional test that measures the maximal distance covered while walking at fast-pace for six minutes
Time Frame: baseline, 8-week
Reporting Status: Not Posted

22. Other Pre Specified Outcome: 7-meter Walk Test [OPTIONAL IN-PERSON VISIT]
Description: functional test that measures comfortable walking speed as participant walks back and forth over 7 meters twice
Time Frame: baseline, 8-week
Reporting Status: Not Posted

23. Other Pre Specified Outcome: Stair Climb Test [OPTIONAL IN-PERSON VISIT]
Description: functional test that measures the time taken to ascend and descend a flight of stairs
Time Frame: baseline, 8-week
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Pressure Pain Threshold [OPTIONAL IN-PERSON VISIT]
Description: a test of pain sensitivity
Time Frame: baseline, 8-week
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Mechanical Temporal Summation [OPTIONAL IN-PERSON VISIT]
Description: a test of central pain sensitization
Time Frame: baseline, 8-week
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Conditioned Pain Modulation [OPTIONAL IN-PERSON VISIT]
Description: a test of descending pain modulation
Time Frame: baseline, 8-week
Reporting Status: Not Posted

27. Other Pre Specified Outcome: Exercise Induced Hypoalgesia [OPTIONAL IN-PERSON VISIT]
Description: a test of change in pain sensitivity after a bout of exercise
Time Frame: baseline, 8-week
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Isometric Knee Extensor Force [OPTIONAL IN-PERSON VISIT]
Description: knee extensor isometric muscle strength
Time Frame: baseline, 8-week
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Isometric Knee Flexor Force [OPTIONAL IN-PERSON VISIT]
Description: knee flexor isometric muscle strength
Time Frame: baseline, 8-week
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Telehealth Usability Questionnaire
Description: scale evaluating the usability and satisfaction of telehealth implementation and services. Each item is rated on a seven-point Likert scale, with a rating of one indicating disagree and a rating of seven indicating agree; higher ratings indicate better system usability
Time Frame: 8-week
Reporting Status: Not Posted

31. Other Pre Specified Outcome: Weekly Log
Description: log of minutes and days spent doing strengthening exercises, aerobic exercises, and mindfulness practice (mindfulness practice only applicable to people in the TMX group). Survey also includes log of oral analgesic use.
Time Frame: Weekly for 14-weeks
Reporting Status: Not Posted

32. Other Pre Specified Outcome: Heal Treatment Expectancy Survey - Short Form
Description: 6-item survey assessing participant's attitude and expectations of the intervention measured on a 5-point likert scale. higher scores indicate more positive attitude and expectations for the treatment
Time Frame: baseline
Reporting Status: Not Posted

33. Other Pre Specified Outcome: Treatment History
Description: a survey that collects information about the treatments the individual has undertaken for their knee osteoarthritis
Time Frame: baseline, week 8, week 14
Reporting Status: Not Posted

34. Other Pre Specified Outcome: eHealth Literacy Scale
Description: 8-item scale measuring one's perceived ability and comfort with accessing digital services for health information. each item is rated on a 5-point likert scale. total scores are summed. higher scores indicate greater perceived skills at using online health information to help solve health problems
Time Frame: baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 14-weeks
Description: The adverse events were self-reported by participants during the course of the study. No serious adverse events were reported by participants in either groups.
Arm/Group | Group TX (Telehealth Exercise) | Group TMX (Telehealth Exercise and Mindfulness)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 8/19 | 3/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group TX (Telehealth Exercise) (N=19) | Group TMX (Telehealth Exercise and Mindfulness) (N=21)
Exacerbation of knee pain (Musculoskeletal and connective tissue disorders) | 4 | 0 — There were four reports of adverse events potentially related to the study in TX group and 0 in the TMX group. These adverse events were related to exacerbation of knee pain. The remaining adverse events were unrelated to the study.
Hernia surgery (Surgical and medical procedures) | 0 | 1 — Adverse event unrelated to study
Flu (Infections and infestations) | 2 | 1 — Adverse event unrelated to study
Ankle injury (Musculoskeletal and connective tissue disorders) | 0 | 1 — Adverse event unrelated to study because event was reported before the start of the intervention sessions
Knee replacement surgery (Surgical and medical procedures) | 1 | 0 — Participant had scheduled a knee replacement surgery during the course of the study
Generally feeling unwell (General disorders) | 1 | 0 — Participant reported generally feeling unwell

LIMITATIONS AND CAVEATS:
There are limitations to consider while interpreting the findings of our study.

1. All outcomes are participant-reported which can introduce bias as we did not include any objective measures (e.g., physical performance).
2. There was lack of diversity in race, education, socioeconomic status, and technological abilities, which limits the external validity of our findings

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-15): https://cdn.clinicaltrials.gov/large-docs/16/NCT05524116/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-05): https://cdn.clinicaltrials.gov/large-docs/16/NCT05524116/ICF_001.pdf